CLINICAL TRIAL: NCT02338505
Title: Teleassisted Surgery for Gynecological Disease in Obese Patients - OB-ALFX
Acronym: OB-ALFX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: SOFAR S.p.A. (Industry)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21264/14
Record Dates: First submitted 2015-01-12; First posted 2015-01-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Benign, Premalignant and Malignant Gynecological Disease Confined to the Pelvis
Keywords: Robotic Surgery; Telelap-ALFX; Gynecological disease
MeSH Terms: conditions — Precancerous Conditions; Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telelap ALF-X in obese patients with gynecological disease (Experimental)
  Interventions: Device: Telelap ALF-X

INTERVENTIONS:
Device: Telelap ALF-X — Patients placed in the dorsal lithotomic position with both legs supported in Allen stirrups with a Trendelenburg tilt. After achieving pneumoperitoneum (12mmHg) through a trans umbilical open access technique, intra-abdominal visualization was obtained with a 10mm 0° HD 3D telescope. During the trocar placement the operative room nurses supported the surgeon in the docking procedures approaching the robotic arms to the operative table, in places established for pelvic surgery. The cockpit is located in one corner of our square shape room; the operative table is surrounded by the three robotic arms unit.
  Through the teleassisted operative ports we could make use of several type of instruments. Movements of both instruments and optic were completely carried out by the surgeon from the cockpit according to the needs of the procedure.
  Other Names: ALF-X teleassisted surgery

SUMMARY:
Phase II prospective single-institutional study.

DETAILED DESCRIPTION:
The aim of this Phase II prospective single-institutional study is to assess feasibility and early complications rate of Telelap ALF-X surgical treatment in obese patients affected by gynecological disease.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* 30 ≤ BMI < 40
* ASA < III
* Ovarian Cyst
* Prophylactic bilateral salpingo-oophorectomy
* Ectopic Pregnancy
* Pelvic Inflammatory Disease
* Sterility/Infertility
* Benign uterine disease (fibromatosis, adenomyosis)
* Endometrial hiperplasia
* Early-stage Endometrial Cancer
* Preneoplastic lesions of the cervix
* IA1 Cervical Cancer
* Pelvic endometriosis

Exclusion Criteria:

* Pregnancy
* Liver disease
* Coagulopathies
* Clinical conditions contraindicating laparoscopy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
intraoperative complication rate | intraoperative
  Operative time, conversion rate, estimated blood loss, visceral injury

SECONDARY OUTCOMES:
postoperative complication rate | 30 days
  Ileus, bleeding, infection/sepsi, thrombosis, rehospitalization, death

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart Rome,, Rome, Rome, Italy

REFERENCES:
- [Result] Gidaro S, Buscarini M, Ruiz E, Stark M, Labruzzo A. Telelap Alf-X: a novel telesurgical system for the 21st century. Surg Technol Int. 2012 Dec;22:20-5. PMID 23225591
- [Result] Gidaro S, Altobelli E, Falavolti C, Bove AM, Ruiz EM, Stark M, Ravasio G, Lazzaretti SS, Maurizio B. Vesicourethral anastomosis using a novel telesurgical system with haptic sensation, the Telelap Alf-X: a pilot study. Surg Technol Int. 2014 Mar;24:35-40. PMID 24706079
- [Result] Lococo A, Larocca V, Marino F, De Filippis AF, Cesario A, Lococo F. Experimental Robotic Pulmonary Lobectomy With the TELELAP/ALFX System in the Ovine Model. Surg Innov. 2015 Jun;22(3):252-6. doi: 10.1177/1553350614549633. Epub 2014 Sep 15. PMID 25225214
- [Result] Falavolti C, Gidaro S, Ruiz E, Altobelli E, Stark M, Ravasio G, Ravasio G, Lazzaretti SS, Buscarini M. Experimental Nephrectomies Using a Novel Telesurgical System: (The Telelap ALF-X)-A Pilot Study. Surg Technol Int. 2014 Nov;25:37-41. PMID 25433265
- See also: Related Info — https://www.policlinicogemelli.it